CLINICAL TRIAL: NCT05847725
Title: Effects of Bandaging and Kinesiotaping® on Pain, Edema, and Functional Level in Patients With Total Knee Arthroplasty in the Early Postoperative Period: A Randomized Clinical Trial
Brief Title: Effects of Bandaging and Kinesiotaping® in Patients With Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gursoy Coskun, Associate Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HU-15/666-21
Record Dates: First submitted 2023-04-01; First posted 2023-05-08 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Knee Osteoarthritis
Keywords: knee arthroplasty; edema; elastic bandages; short stretch bandages; kinesio tape
MeSH Terms: conditions — Osteoarthritis, Knee; Edema

STUDY DESIGN:
Intervention Model Description: The study included a three parallel group of blinded evaluators. These cases were followed up with a planned follow-up program between preoperative and postoperative three months.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Elastic bandaging (Experimental): Patients who have undergone TKA for primary knee OA
  Interventions: Other: Elastic bandaging
- Short stretch bandaging (Experimental): Patients who have undergone TKA for primary knee OA
  Interventions: Other: Short stretch bandaging
- Kinesio taping (Experimental): Patients who have undergone TKA for primary knee OA
  Interventions: Other: Kinesio taping

INTERVENTIONS:
Other: Elastic bandaging — The bandages were wrapped circularly along the extremity from the toes to the groin, drawing an "8" at the ankle with a 50% overlap rate, starting with 80% tension and decreasing the pressure proximally.
  Arms: Elastic bandaging
Other: Short stretch bandaging — Short tension bandage application was started on postoperative day 1 following the removal of the drains. According to the width of the extremity, using short tension bandages of 6, 8 and 10 cm width, starting from the sole of the foot, the first layer was wrapped circularly with 50% overlapping rate, 80% tension, and wrapped from the sole of the foot to the groin.
  Arms: Short stretch bandaging
Other: Kinesio taping — Kinesio taping was applied in the form of a fan by cutting into 4 longitudinal pieces using the lymphatic correction technique with 15-20% tension, starting from the periphery of the inguinal lymph nodes on the medial, anterior and lateral of the leg, following the removal of the drains from the 1st post-op day.
  Arms: Kinesio taping

SUMMARY:
The study aimed to compare the effectiveness of elastic bandaging, Kinesio taping, and short stretch bandaging techniques on postoperative pain, edema, and functional level in the early stage after total knee arthroplasty.

DETAILED DESCRIPTION:
The study was conducted on 30 volunteer subjects who underwent unilateral total knee arthroplasty surgery. Thirty participants who underwent unilateral total knee arthroplasty were divided into the Elastic Bandage Group (n=10), Kinesio Tape group (n=10), and Short Stretch Bandage group (n=10). All treatments were stopped on the eighth day. All measurements taken preoperatively were repeated postoperative 1st, 3rd, 5th, 8th, 14th, 28th days, 6th week, and 3rd month. The functional level was measured in the sixth week and third month.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older patients who had undergone unilateral TKA surgery for primary knee osteoarthritis, rheumatoid arthritis, and posttraumatic arthritis.

Exclusion Criteria:

* Body mass index greater than or equal to 35 kg/m2,
* Having a neurological or peripheral vascular disease,
* Having a contraindication condition for compression application (e.g., acute cellulitis, arterial insufficiency, unstable heart disease, acute deep vein thrombosis), and kinesio taping application (e.g., presence of active infectious, lymphedema and/ or cancer history)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | up to sixth weeks
  Pain intensity, Minumum score 0: no pain, maximum score 10: worst pain

SECONDARY OUTCOMES:
Measuring Tape Measure | up to sixth weeks
  Edema
The Knee Society Clinical Scoring System | up to sixth weeks
  Functional level assessment, maximum score 100, <60 poor, 60-69 average, 70-84 good, 85-100 excellent

CONTACTS AND LOCATIONS:
Overall Officials: Gürsoy Coşkun, Assoc. Prof, Principal Investigator — Hacettepe University